CLINICAL TRIAL: NCT05422430
Title: Effect of Rebreathing-induced Hypoxia on the Response to an Oral Glucose Tolerance Test
Brief Title: Rebreathing-induced Hypoxia and Glucose Levels
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Sophie Lalande, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001555
Record Dates: First submitted 2022-05-08; First posted 2022-06-16 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous breathing (Sham Comparator): Participants will be spontaneously breathing during an oral glucose tolerance test.
  Interventions: Behavioral: Spontaneous breathing
- Rebreathing-induced hypoxia (Experimental): Participants will rebreathe room air from a low-volume closed-circuit system for a period of 2 minutes.
  Interventions: Behavioral: Rebreathing-induced hypoxia

INTERVENTIONS:
Behavioral: Rebreathing-induced hypoxia — Participants will rebreathe room air from a low-volume closed-circuit system for a period of 2 minutes.
  Arms: Rebreathing-induced hypoxia
Behavioral: Spontaneous breathing — Participants will be spontaneously breathing during an oral glucose tolerance test.
  Arms: Spontaneous breathing

SUMMARY:
The aim of this research project is to determine the effect of repeated maximal voluntary apneas on glucose uptake during an oral glucose tolerance test in healthy individuals, individuals with prediabetes and patients with type 2 diabetes.

DETAILED DESCRIPTION:
It is predicted that 1 in 3 adults will develop diabetes by 2050, implying that a large percentage of the population will become at high risk for cardiovascular disease, the most common cause of death in patients with type 2 diabetes. While regular exercise reduces insulin resistance and the elevated glucose levels associated with type 2 diabetes, only 28% of the adult population with diabetes meet physical activity recommendations. There is therefore an urgent need to identify alternative, non-pharmacological interventions that prevent and treat type 2 diabetes.

A reduced oxygen availability, or hypoxia, is widely implicated in the development of insulin resistance. Paradoxically, hypoxia also triggers glucose uptake independently from the actions of insulin. Indeed, breathing low levels of oxygen stimulates glucose uptake in skeletal muscles by activating 5' adenosine monophosphate-activated protein kinase (AMPK). Discrepancies on the effect of hypoxia on glucose homeostasis may be attributed to the duration and type (nocturnal vs. diurnal) of hypoxic exposure. For example, the many severe hypoxic bouts associated with obstructive sleep apnea are associated with a worsened glycemic control while hypoxic exposure consisting of a limited number of short bouts of moderate hypoxia improves glycemic control. Therefore, an intervention that can induce brief hypoxic conditions, as observed through a reduced fraction of inspired oxygen, could attenuate the postprandial increase in glucose levels.

Fraction of inspired oxygen can be reduced by rebreathing into a low-volume closed-circuit system containing ambient air for few minutes. Thus, the aim of this research project is to determine the effect of few bouts of rebreathing-induced hypoxia on glucose uptake during an oral glucose tolerance test in healthy individuals, individuals with prediabetes and patients with type 2 diabetes. If our expected outcomes are met, our next step will be to determine whether repeated sessions of rebreathing-induced hypoxia (5 sessions per week over 1-3 months) results in improvements in glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years old

Exclusion Criteria:

* Have uncontrolled stage 2 hypertension (˃140/90 mmHg)
* Are smokers
* Are pregnant
* Have a history of cardiovascular disease or indication of cardiovascular disease such as myocardial infarction, left ventricular hypertrophy, ischemic heart disease (or prior ischemia), stroke, and/or other vascular disease
* Have a history of lung disease
* Are taking insulin or more than one antihypertensive medication
* Have poorly controlled diabetes: HbA1c levels ˃ 9%
* Have been previously diagnosed with diabetic complications (nephropathy, neuropathy, retinopathy) by their family doctor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in plasma glucose levels | Collected at min 0, 30, 60, 90 and 120 minutes of the oral glucose tolerance test
  Plasma glucose levels obtained from a venous catheter during a 2-hour oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lalande, Principal Investigator — UT Austin
Locations (1):
- The Unviersity of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Background] Boyle JP, Thompson TJ, Gregg EW, Barker LE, Williamson DF. Projection of the year 2050 burden of diabetes in the US adult population: dynamic modeling of incidence, mortality, and prediabetes prevalence. Popul Health Metr. 2010 Oct 22;8:29. doi: 10.1186/1478-7954-8-29. PMID 20969750
- [Background] Resnick HE, Foster GL, Bardsley J, Ratner RE. Achievement of American Diabetes Association clinical practice recommendations among U.S. adults with diabetes, 1999-2002: the National Health and Nutrition Examination Survey. Diabetes Care. 2006 Mar;29(3):531-7. doi: 10.2337/diacare.29.03.06.dc05-1254. PMID 16505501
- [Background] Azevedo JL Jr, Carey JO, Pories WJ, Morris PG, Dohm GL. Hypoxia stimulates glucose transport in insulin-resistant human skeletal muscle. Diabetes. 1995 Jun;44(6):695-8. doi: 10.2337/diab.44.6.695. PMID 7789635
- [Background] Cartee GD, Douen AG, Ramlal T, Klip A, Holloszy JO. Stimulation of glucose transport in skeletal muscle by hypoxia. J Appl Physiol (1985). 1991 Apr;70(4):1593-600. doi: 10.1152/jappl.1991.70.4.1593. PMID 2055841
- [Background] Mu J, Brozinick JT Jr, Valladares O, Bucan M, Birnbaum MJ. A role for AMP-activated protein kinase in contraction- and hypoxia-regulated glucose transport in skeletal muscle. Mol Cell. 2001 May;7(5):1085-94. doi: 10.1016/s1097-2765(01)00251-9. PMID 11389854
- [Background] Louis M, Punjabi NM. Effects of acute intermittent hypoxia on glucose metabolism in awake healthy volunteers. J Appl Physiol (1985). 2009 May;106(5):1538-44. doi: 10.1152/japplphysiol.91523.2008. Epub 2009 Mar 5. PMID 19265062
- [Background] Newhouse LP, Joyner MJ, Curry TB, Laurenti MC, Man CD, Cobelli C, Vella A, Limberg JK. Three hours of intermittent hypoxia increases circulating glucose levels in healthy adults. Physiol Rep. 2017 Jan;5(1):e13106. doi: 10.14814/phy2.13106. Epub 2017 Jan 13. PMID 28087818
- [Background] Duennwald T, Gatterer H, Groop PH, Burtscher M, Bernardi L. Effects of a single bout of interval hypoxia on cardiorespiratory control and blood glucose in patients with type 2 diabetes. Diabetes Care. 2013 Aug;36(8):2183-9. doi: 10.2337/dc12-2113. Epub 2013 Mar 27. PMID 23536585
- [Background] Costalat G, Lemaitre F, Tobin B, Renshaw G. Intermittent hypoxia revisited: a promising non-pharmaceutical strategy to reduce cardio-metabolic risk factors? Sleep Breath. 2018 Mar;22(1):267-271. doi: 10.1007/s11325-017-1459-8. Epub 2017 Feb 2. PMID 28155101
- [Background] de Bruijn R, Richardson M, Schagatay E. Increased erythropoietin concentration after repeated apneas in humans. Eur J Appl Physiol. 2008 Mar;102(5):609-13. doi: 10.1007/s00421-007-0639-9. Epub 2007 Dec 19. PMID 18097682